CLINICAL TRIAL: NCT04977583
Title: The Effect of Screening and Referral for Social Determinants of Health on Veterans' Outcomes
Brief Title: Unmet Social Needs Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency); Ralph H. Johnson VA Medical Center (U.S. Federal Agency); Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IIR 19-013
Record Dates: First submitted 2021-07-16; First posted 2021-07-27 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Disease; Hypertension; Diabetes Mellitus; Hyperlipidemia
Keywords: Social Determinants of Health; Veterans; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Diabetes Mellitus; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: The investigators are implementing a three-armed randomized controlled trial (RCT) at three VA sites to compare outcomes among Veterans with one or more unmet social needs randomized within each site to one of three intervention arms. The investigators have the following study arms/conditions: unmet needs screening only by Research Assistant ("Screening" arm"; Screening plus provision of a tailored Resource Sheet listing available resources to address identified needs ("Awareness" arm); Screening plus provision of tailored Resource Sheet plus research team social worker-supported referral to assist with connection to resources to address unmet needs ("Assistance" arm).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Screening (Experimental): Participants in this arm will be screened for unmet social needs and receive a post card that includes a list of generic VA crisis and homeless hotlines.
  Interventions: Behavioral: Unmet Need Screening
- Awareness (Experimental): Participants in this arm will be screened for unmet social needs, receive a post card that includes a list of generic VA crisis and homeless hotlines, and receive a Resource Sheet tailored to the unmet needs identified in the unmet need screen. The Resource Sheet will include the names of available resources within the VA and/or local community that can help to address the identified need(s) and contact information and hours of operation.
  Interventions: Behavioral: Unmet Need Screening; Behavioral: Unmet Need Referral - Resource Sheet
- Assistance (Experimental): Participants in this arm will be screened for unmet social needs, receive a post card that includes a list of generic VA crisis and homeless hotlines, receive a tailored Resource Sheet, and be offered assistance from a Social Worker. If accepted, the SW will contact the participant and work with them over a period of 8 weeks to help facilitate their connection to resources than can help to address the unmet need(s) identified in the unmet need screen.
  Interventions: Behavioral: Unmet Need Screening; Behavioral: Unmet Need Referral - Resource Sheet; Behavioral: Unmet Need Referral Assistance

INTERVENTIONS:
Behavioral: Unmet Need Screening — Participants are screened by phone for unmet social needs (e.g., utility insecurity, social isolation), hereafter referred to as the "index screen". The index screen occurs prior to randomization.
Behavioral: Unmet Need Referral - Resource Sheet — Participants receive a Resource Sheet(s) tailored to the unmet need(s) identified in the index screen. For each unmet need, a Resource Sheet will include the names of available resource within the VA and/or the local community that can help address the unmet need and contact information (address, phone, website, email) and hours of operation.
  Arms: Assistance; Awareness
Behavioral: Unmet Need Referral Assistance — Participants receive assistance from a Social Worker (SW) to facilitate connection to resources that can help to address unmet need(s) identified in the index screen. Assistance includes 1) conducting a standardized bio-psychosocial assessment; 2) motivational interviewing methods to uncover details of the Veteran's unmet needs and identify barriers to resolving the unmet needs, and; 3) developing an action plan for the Veteran to connect with resources and address needs. The SW will conduct initial follow-up by phone one week after the interview/action plan development, with planned subsequent phone outreach every two weeks for up to seven weeks.
  Arms: Assistance

SUMMARY:
The impacts of unmet social needs, such as homelessness, inconsistent access to food, and exposure to violence on health are well-established, especially for cardiovascular disease. A limited but growing body of evidence suggests that screening for and addressing these needs - also referred as social determinants of health -- in clinic settings helps to connect patients to resources to address unmet needs and has the potential to improve health outcomes. Veterans carry a high burden of unmet needs. At present, VA systematically screens for only two unmet needs; homelessness and food insecurity. The investigators propose to assess the efficacy of systematically screening Veterans for nine unmet needs (i.e., housing, food insecurity, utility insecurity, transportation, legal problems, employment, safety, stress, and social isolation), and compare the effect of referral mechanisms of varying intensity on Veterans' connection to resources, reduction of unmet needs, treatment adherence, reduced preventable hospitalizations, and clinical outcomes.

DETAILED DESCRIPTION:
Background: Despite medical advances, up to 70% of health outcomes are due to social determinants of health (SDoH) - the conditions in which people live and work that shape whether basic needs (e.g., housing, food) are met. These associations are especially well documented for cardiovascular disease (CVD). In response, health policy leaders recommend screening and referral (S&R) for unmet needs in clinical settings, and the American Heart Association recently concluded that the most significant opportunities for reducing CVD death and disability lie with addressing the social determinants of cardiovascular outcomes. A limited but promising evidence base supports these recommendations but more rigorous research is needed to guide how best to intervene on unmet needs that affect health.

Significance/Impact: This project addresses the Office of Social Work's priority to link Veterans with resources and services in support of treatment goals, the Office of Patient Centered Care and Cultural Transformation's priority to enhance the physical, emotional, and social well-being of the whole person, the Office of Health Equity's priority to reduce disparities, and the HSR&D priorities of health equity and population health. Our study will provide much-needed evidence to document the burden of Veterans' unmet needs, inform how best to address unmet needs, and assess how such a process can affect adherence (to medications and appointments), utilization, and clinical outcomes.

Innovation: VA currently systematically screens for only two unmet needs (homelessness and food insecurity). Identification of other unmet needs (and referral to address them) occurs on an ad hoc basis, with varying approaches among clinics/ clinicians. The investigators will implement comprehensive screening of eight unmet needs and systematic referral, developing tools and processes that, if efficacious, can be implemented within VA (and other) clinical systems. VA is currently funding several studies related to SDoH, but none test interventions that systematically identify a wide range of unmet social needs among Veterans and connect Veterans with identified needs to social service resources.

Specific Aims: 1) Describe the burden and distribution of nine unmet needs (i.e., housing; food insecurity; utility insecurity; transportation; legal guidance; employment; safety; and social isolation) among Veterans with or at-risk for CVD, and identify their associations with sociodemographic characteristics, and baseline health-related behaviors and clinical outcomes; 2) Compare the effects of three S&R study intervention conditions of varying intensity on Veterans' connection to new SDoH resources (primary outcome), reduction of unmet needs, adherence, and clinical outcomes, and 3) Identify barriers and facilitators to Veterans' connecting with social services and having needs met, and explanatory factors for observed RCT outcomes.

Methodology: The investigators propose a 3-year, two-phased mixed methods study. In Phase One (Aims 1 and 2), the investigators will implement a three-armed randomized controlled trial at three VA sites to compare outcomes among Veterans randomized within each site to one of three study conditions: screening only; screening plus provision of tailored resource sheets; or screening plus resource sheets plus social work support. For each Veteran, the investigators will examine associations of unmet needs with baseline outcomes (Aim 1), and longitudinally examine the impact of each approach on connection to new SDoH resources and follow-up outcomes over a 12-month period (Aim 2). In Phase Two (Aim 3), the investigators will conduct interviews with Veterans and representatives of the VA- and community-based programs to which Veterans are referred because of the trial to identify facilitators and barriers and potential explanatory factors related to the relative success of the interventions.

Implementation/Next Steps: If the intervention yields positive results, findings will be used by partners to support more widespread implementation of it throughout VA.

ELIGIBILITY:
Inclusion Criteria:

* Veterans enrolled in one of three VA medical centers:

  * 1) VA Boston Healthcare System
  * 2) Corporal Michael J. Crescenz VA Medical Center (Philadelphia)
  * 2) Ralph H. Johnson VA Medical Center (Charleston)
* Veterans with, or at risk for, cardiovascular disease (CVD) who had at least 1 PC visit in the prior year
* CVD patients are defined as those with International Classification of Disease 10 (ICD10) diagnoses indicating:

  * coronary artery disease
  * cerebrovascular disease
  * peripheral artery disease
* Patients at-risk for CVD are defined as having diagnoses of hypertension, diabetes mellitus (DM), or hyperlipidemia

Exclusion Criteria:

* Impaired decision-making
* Illiterate or have limited or no English proficiency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Gurewich, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (3):
- United States (3):
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share final quantitative data sets underlying all publications resulting from the proposed research, after deidentification. A limited data set will be created and shared pursuant to a Data Use Agreement appropriately limiting use if the data set and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or reidentify) any individual whose data are included in the dataset. Prior to distribution, a local privacy officer will certify that the all datasets contain no protected health information. The PI will maintain a crosswalk between the analytical data set(s) and the public release data sets so that a VA-approved auditor or the PI could conduct or facilitate validation if needed. Qualitative data will not be shared. The sensitive nature of the study data precludes asking participants to consent and grant HIPAA authorization for sharing.
Supporting Information: Study Protocol
Time Frame: Quantitative data meeting VA standards for disclosure to the public will be made available within one year of publication. The quantitative analytical datasets and statistical code used in the publication will be retained for 6 years, in accordance with VA record retention policy.
Access Criteria: Quantitative data sets will be made available to investigators whose proposed use of the data have been approved by an independent review committee identified for that purpose. The proposed analyses must be for individual participant data meta-analysis.

REFERENCES:
- [Result] Gurewich D, Kressin N, Bokhour BG, Linsky AM, Dichter ME, Hunt KJ, Fix GM, Niles BL. Randomised controlled trial evaluating the effects of screening and referral for social determinants of health on Veterans' outcomes: protocol. BMJ Open. 2022 Sep 23;12(9):e058972. doi: 10.1136/bmjopen-2021-058972. PMID 36153033
- [Derived] Gurewich D, Hunt K, Bokhour B, Fix G, Friedman H, Li M, Linsky AM, Niles B, Dichter M. Screening and Referral for Social Needs Among Veterans: A Randomized Controlled Trial. J Gen Intern Med. 2025 Aug;40(11):2732-2739. doi: 10.1007/s11606-024-09105-x. Epub 2025 Jan 23. PMID 39849274

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from April 2022 - June 2023. Trained research assistants (RAs) recruited participants by phone.
Pre-assignment Details: Participants needed to screen positive for one of nine needs to be assigned to an arm. Participants with zero needs were not eligible for the trial and thus not randomized to an arm.
Groups:
- Assistance: Participants in this arm will receive the same interventions as Arm 2 (screened by phone for unmet social needs, receive post card listing generic resources, and receive tailored resource sheets) plus be offered assistance from a Social Worker. If accepted, the SW will contact the participant and work with them over a period of 8 weeks to help facilitate their connection to resources than can help to address the unmet need(s) identified in the unmet need screen.
  Unmet Need Screening: Participants are screened by phone for unmet social needs (e.g., utility insecurity, social isolation), hereafter referred to as the "index screen". The index screen occurs prior to randomization.
  Unmet Need Referral - Resource Sheet: Participants receive a Resource Sheet(s) tailored to the unmet need(s) identified in the index screen. For each unmet need, a Resource Sheet will include the names of available resource within the VA and/or the local community that can help address the unmet need and contact information (address, phone, website, email) and hours of operation.
Period: Overall Study
Arm/Group | Screening | Awareness | Assistance
Started | 161 | 160 | 158
8 Week Screen | 143 | 141 | 133
6 Month Screen | 135 | 133 | 138
Completed | 150 | 154 | 144
Not Completed | 11 | 6 | 14
Not completed — Lost to Follow-up | 8 | 4 | 13
Not completed — Withdrawal by Subject | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Screening | Awareness | Assistance | Total
Number analyzed (Participants) | 161 | 160 | 158 | 479
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.58 (11.55) | 63.96 (12.17) | 64.16 (11.50) | 64.24 (11.72)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Women | 12 | 10 | 21 | 43
  Gender: Men | 148 | 150 | 137 | 435
  Gender: Transgender Women | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 10 | 9 | 30
  Not Hispanic or Latino | 150 | 150 | 149 | 449
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 1 | 4
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 87 | 70 | 72 | 229
  White | 74 | 84 | 80 | 238
  More than one race | 0 | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 1 | 1
Baseline Average Needs per Participant [Mean (Standard Deviation); unit: Count of social needs] — All study participants were surveyed by phone at enrollment. The survey screened participants for 9 social needs (food, housing, legal, utilities, social disconnection, transportation, stress, exposure to violence, employment). Survey measures were based on existing social need screens. The baseline measure was based on a count of needs that each participant identified at the index screen.
  Count of social needs | 2.45 (1.36) | 2.53 (1.61) | 2.54 (1.39) | 2.51 (1.45)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Connected With a New Resource
Description: Defined as participant connecting to one or more resources since the index unmet need screen and assessed via a participant survey administered 8 weeks following the index unmet need screen. The survey will ask: "Since you completed the unmet social need screen on (insert date), were you able to connect with any of the programs or resources for help with (insert need(s) identified)".
Time Frame: 8 weeks
Population: One participant in arm 3 was excluded from analysis due to missing race information.
Measure: Count of Participants; unit: Participants
Arm/Group | Screening | Awareness | Assistance
Number analyzed (Participants) | 161 | 160 | 157
Participants | 40 | 41 | 51
Statistical Analysis 1: Comparison: Screening; This test is comparing Arm 1 (screening) to Arm 2 (awareness); Test type: Superiority; p = 0.6243, Mixed Models Analysis; Odds Ratio (OR) = 1.138, 95% CI 2-sided [0.679 to 1.904], Standard Error of Mean 0.2625
Statistical Analysis 2: Comparison: Screening; This test compares Arm 1 (screening) to arm 3 (assistance); Test type: Superiority; p = 0.1146, Mixed Models Analysis; Odds Ratio (OR) = 1.497, 95% CI 2-sided [0.908 to 2.469], Standard Error of Mean 0.2553

2. Primary Outcome: Mean Count of Resources Connected To
Description: Defined as a count of resources that a participant connected to since the index unmet need screen and assessed via a participant survey administered 8 weeks following the index unmet need screen. The survey will ask: "Since you completed the unmet social need screen on (insert date), were you able to connect with any of the programs or resources for help with (insert need(s) identified)".
Time Frame: 8 weeks
Population: One participant in arm 3 was excluded from analysis due to missing race information.
Measure: Mean (Standard Deviation); unit: Count of resources connected
Arm/Group | Screening | Awareness | Assistance
Number analyzed (Participants) | 161 | 160 | 157
Count of resources connected | 0.40 (.79) | 0.40 (0.83) | 0.47 (0.77)
Statistical Analysis 1: Comparison: Screening; This test is comparing Arm 1 (screening) to Arm 2 (awareness); Test type: Superiority; p = 0.856, Poisson; We used total needs as an offset; Risk Ratio (RR) = 0.963, 95% CI 2-sided [0.641 to 1.447], Standard Error of Mean 0.2078
Statistical Analysis 2: Comparison: Screening; This test is comparing Arm 1 (screening) to Arm 3 (assistance); Test type: Superiority; p = 0.5248, Poisson; Risk Ratio (RR) = 1.136, 95% CI 2-sided [0.768 to 1.681], Standard Error of Mean 0.1999

3. Secondary Outcome: Unmet Need Reduction - Any
Description: The investigators will compare the results from the index screen for unmet needs to those from the unmet needs screen administered six months after the index screen. The investigators will define unmet need reduction in two ways. This measure is one or more of baseline unmet needs no longer identified as an unmet need at the 6-month rescreen.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Screening | Awareness | Assistance
Number analyzed (Participants) | 161 | 160 | 158
Participants | 82 | 73 | 74
Statistical Analysis 1: Comparison: Screening; This is Arm 1 compared to Arm 2; Test type: Superiority; p = .5582, Regression, Logistic; Odds Ratio (OR) = 0.866, 95% CI 2-sided [0.536 to 1.400], Standard Error of Mean 0.220
Statistical Analysis 2: Comparison: Screening; This is Arm 1 compared to Arm 3; Test type: Superiority; p = 0.5196, Regression, Logistic; Odds Ratio (OR) = 0.854, 95% CI 2-sided [0.528 to 1.381], Standard Error of Mean 0.217

4. Secondary Outcome: Emergent Visits (Urgent Care and Emergency Department Visits)
Description: The measure is change in Emergency Department and urgent care visits. Change is calculated as (mean at 12 months - mean at baseline). The investigators will assess this measure using CDW.
Time Frame: 12 months compared to baseline
Measure: Mean (Standard Deviation); unit: Mean difference in emergent visits
Arm/Group | Screening | Awareness | Assistance
Number analyzed (Participants) | 161 | 160 | 158
Mean difference in emergent visits | 0.19 (2.36) | 0.53 (2.64) | -0.01 (2.15)
Statistical Analysis 1: Comparison: Screening; This is arm 1 compared to arm 2; Test type: Superiority; p = 0.2105, ANOVA; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.821 to 2.454], Standard Error of Mean .2794
Statistical Analysis 2: Comparison: Screening; This is arm 1 compared to arm 3; Test type: Superiority; p = .4143, ANOVA; Odds Ratio (OR) = 0.7944, 95% CI 2-sided [0.4574 to 1.379], Standard Error of Mean 0.2816

5. Secondary Outcome: Medication Adherence
Description: The investigators will assess adherence to CVD and CVD risk factor medications, including all possible drug class codes (CV000-CV900, encompassing Antilipemic agents and antihypertensives for the subsets of patients prescribed these medications) and, among the subset of patients with DM, diabetes medications (HS501-509). The measure will be based on pharmacy dispensing data from CDW to specify the proportion of days covered (PDC) of each medication. To calculate this, the investigators will count the # of days dispensed in relation to the dispensing period. The numerator will be based on the prescription fill dates and # of days dispensed to determine the number of outpatient days for which each medication was supplied. Patients will be considered adherent if they achieved a PDC > 80%. The measure is change in medication adherence. Change is calculated as (mean at 12 months - mean at baseline). The investigators will assess this measure using CDW.
Time Frame: 12 months compared to baseline
Measure: Mean (Standard Deviation); unit: med adherence% post - med adherence% pre
Arm/Group | Screening | Awareness | Assistance
Number analyzed (Participants) | 161 | 160 | 158
med adherence% post - med adherence% pre | 0.01 (0.15) | 0.01 (0.12) | 0.03 (0.13)
Statistical Analysis 1: Comparison: Screening; This arm 1 compared to arm 2; Test type: Superiority; p = 0.9775, ANOVA; Odds Ratio (OR) = 0.9995, 95% CI 2-sided [0.9665 to 1.0336], Standard Error of Mean 0.0171
Statistical Analysis 2: Comparison: Screening; This arm 1 compared to arm 3; Test type: Superiority; p = 0.3194, ANOVA; Odds Ratio (OR) = 1.017, 95% CI 2-sided [0.9832 to 1.0534], Standard Error of Mean 0.0176

6. Secondary Outcome: Clinic Visit Appointment Attendance ("No-show")
Description: For each patient, the investigators will calculate a no-show rate, or the proportion of primary care and cardiology appointments that are classified as no-show, relative to the total number of appointments scheduled in both, following the approach taken by other VA investigators using CDW data to assess this metric. The numerator ("no-shows") consists of appointments marked as a no-show and appointments canceled by the patient or clinic after the appointment time. The denominator ("total appointments") consists of no-shows and completed appointments. The measure is change in no shows. Change is calculated as (mean at 12 months - mean at baseline). The investigators will assess this measure using CDW.
Time Frame: 12 months compared to baseline
Measure: Mean (Standard Deviation); unit: Number of appointments missed
Arm/Group | Screening | Awareness | Assistance
Number analyzed (Participants) | 161 | 160 | 158
Number of appointments missed | -0.14 (1.52) | -0.06 (1.40) | 0.22 (1.27)
Statistical Analysis 1: Comparison: Screening; This is arm 1 compared to arm 2; Test type: Superiority; p = 0.8623, ANOVA; Odds Ratio (OR) = 1.0284, 95% CI 2-sided [0.7497 to 1.4107], Standard Error of Mean 0.1613
Statistical Analysis 2: Comparison: Screening; This is arm 1 compared to arm 3; Test type: Superiority; p = 0.0534, ANOVA; Odds Ratio (OR) = 1.3701, 95% CI 2-sided [0.9962 to 1.8844], Standard Error of Mean 0.1626

7. Secondary Outcome: Systolic Blood Pressure (BP)
Description: BP is measured at every PC visit, and the investigators will obtain these measurements from CDW. In the rare case of missing BP data, the investigators will exclude such Veterans from the analysis. Because BP outcomes are also affected by clinicians' adjustment or titration of antihypertensive medications, the investigators will assess the effects of controlling for treatment intensification (TI), using methods similar to the published approaches used in prior work. The investigators will use the following formula to measure TI: (visits with medication changes-visits with elevated BP) / (number of clinic visits).
Time Frame: 12 months compared to baseline
Measure: Mean (Standard Deviation); unit: Mean change in mmHg
Arm/Group | Screening | Awareness | Assistance
Number analyzed (Participants) | 161 | 160 | 158
Mean change in mmHg | -1.20 (9.37) | -0.27 (12.80) | -0.23 (13.61)
Statistical Analysis 1: Comparison: Screening; This is arm 1 compared to arm 2; Test type: Superiority; p = 0.5701, ANOVA; Odds Ratio (OR) = 2.298, 95% CI 2-sided [0.1304 to 40.5121], Standard Error of Mean 1.4640
Statistical Analysis 2: Comparison: Screening; This is arm 1 compared to arm 3; Test type: Superiority; p = 0.3016, ANOVA; Odds Ratio (OR) = 4.560, 95% CI 2-sided [0.2571 to 80.8746], Standard Error of Mean 1.467

8. Secondary Outcome: Hemoglobin A1c (HbA1c)
Description: HbA1c is available from CDW. The investigators anticipate approximately 40% of our RCT sample to have DM, based on a preparatory-to-research analysis of CDW data. To ensure the values reflect health status around the time of the index screen and the 6 and 12-month follow-up window, the investigators will only include Veterans with DM who have an Hba1c in the 6 months prior to each time point. Approximately 17% of patients with DM do not have an HbA1c test within VA in the prior year.
Time Frame: 12 months compared to baseline
Population: This only contains people who are indicated as having diabetes
Measure: Mean (Standard Deviation); unit: Mean % glycated hemoglobin
Arm/Group | Screening | Awareness | Assistance
Number analyzed (Participants) | 75 | 81 | 52
Mean % glycated hemoglobin | -0.42 (1.11) | -0.03 (1.43) | 0.11 (1.12)
Statistical Analysis 1: Comparison: Screening; This is arm 1 compared to arm 2; Test type: Superiority; p = 0.0870, ANOVA; Odds Ratio (OR) = 1.522, 95% CI 2-sided [0.944 to 2.454], Standard Error of Mean 0.2438
Statistical Analysis 2: Comparison: Screening; This is arm 1 compared to arm 3; Test type: Superiority; p = 0.0354, ANOVA; Odds Ratio (OR) = 1.850, 95% CI 2-sided [1.048 to 3.264], Standard Error of Mean 0.2897

9. Secondary Outcome: Unmet Need Reduction - Percent
Description: The investigators will compare the results from the index screen for unmet needs to those from the unmet needs screen administered six months after the index screen. The investigators will define unmet need reduction in two ways. This measure is percentage of baseline needs not reported as unmet needs at 6-month rescreen.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Percent of Needs not reported as unmet
Arm/Group | Screening | Awareness | Assistance
Number analyzed (Participants) | 161 | 160 | 158
Percent of Needs not reported as unmet | 30.37 (36.6) | 27.11 (35.98) | 27.88 (35.91)
Statistical Analysis 1: Comparison: Screening; This is arm 1 compared to arm 2; Test type: Superiority; p = 0.3063, ANOVA; Odds Ratio (OR) = 0.618, 95% CI 2-sided [0.246 to 1.553], Standard Error of Mean 0.333
Statistical Analysis 2: Comparison: Screening; This is arm 1 compared to arm 3; Test type: Superiority; p = .4378, ANOVA; Odds Ratio (OR) = .679, 95% CI 2-sided [.256 to 1.803], Standard Error of Mean 0.3946

10. Secondary Outcome: Diastolic Blood Pressure (BP)
Description: as for outcome 7
Time Frame: 12 months compared to baseline
Measure: Mean (Standard Deviation); unit: Mean change in mmHg
Arm/Group | Screening | Awareness | Assistance
Number analyzed (Participants) | 161 | 160 | 158
Mean change in mmHg | -0.43 (6.11) | -1.17 (7.07) | -0.11 (7.44)
Statistical Analysis 1: Comparison: Screening; This is arm 1 compared to arm 2; Test type: Superiority; p = 0.4134, ANOVA; Odds Ratio (OR) = 0.5083, 95% CI 2-sided [0.1006 to 2.5687], Standard Error of Mean 0.8265
Statistical Analysis 2: Comparison: Screening; This is arm 1 compared to arm 3; Test type: Superiority; p = 0.4705, ANOVA; Odds Ratio (OR) = 1.819, 95% CI 2-sided [0.3588 to 9.2230], Standard Error of Mean 0.8283

11. Post Hoc Outcome: Number of Participants Who Connected With a New Resource (With Arm 3 Refusals Removed)
Description: as for outcome 1
Time Frame: 8 weeks
Population: Participants in arm 3 could refuse to speak with a social worker. This analysis is with arm 3 refusals removed. The participant with no race info refused arm 3 and is excluded from the 125.
Measure: Count of Participants; unit: Participants
Arm/Group | Screening | Awareness | Assistance
Number analyzed (Participants) | 161 | 160 | 125
Participants | 40 | 41 | 44
Statistical Analysis 1: Comparison: Screening; Test type: Superiority; p = 0.0347, Mixed Models Analysis; Odds Ratio (OR) = 1.765, 95% CI 2-sided [1.044 to 2.987], Standard Error of Mean 0.2684 — This analysis is arm 1 compared to arm 3. Arm 3 is the numerator and arm 1 is the denominator

12. Post Hoc Outcome: Number of Participants Who Connected With a New Resource (Elixhauser Score >=4 Only)
Description: Defined as participant connecting to one or more resources since the index unmet need screen and assessed via a participant survey administered 8 weeks following the index unmet need screen. The survey will ask: "Since you completed the unmet social need screen on (insert date), were you able to connect with any of the programs or resources for help with (insert need(s) identified)". This was an ad-hoc sub-group analysis consisting of Veterans with an Elixhauser score of 4 or greater. The Elixhauser comorbidity index is a measure of comorbidity based on ICD-10 codes. A higher number indicates more comorbidities. The scale is 0-30.
Time Frame: 8 weeks
Population: Elixhauser score >=4 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Screening | Awareness | Assistance
Number analyzed (Participants) | 96 | 89 | 79
Participants | 21 | 23 | 31
Statistical Analysis 1: Comparison: Screening; Test type: Superiority; p = 0.1160, Mixed Models Analysis; Odds Ratio (OR) = 1.734, 95% CI 2-sided [0.875 to 3.436], Standard Error of Mean 0.3489 — This analysis compares arm 1 to arm 2. Arm 2 is the numerator and Arm 1 is the denominator
Statistical Analysis 2: Comparison: Screening; Test type: Superiority; p = 0.0134, Mixed Models Analysis; Odds Ratio (OR) = 2.376, 95% CI 2-sided [1.202 to 4.695], Standard Error of Mean 0.3475

13. Post Hoc Outcome: Number of Participants Who Connected With a New Resource (VA Priority Groups 4 & 5 Only)
Description: Defined as participant connecting to one or more resources since the index unmet need screen and assessed via a participant survey administered 8 weeks following the index unmet need screen. The survey will ask: "Since you completed the unmet social need screen on (insert date), were you able to connect with any of the programs or resources for help with (insert need(s) identified)". This was an ad-hoc sub-group analysis consisting of Veterans in VA priority groups 4 & 5 (of which 95% of Veterans were in priority group 5). Veterans applying for VHA healthcare are assigned to one of eight priority groups based on eligibility criteria including income and service connected disability. A lower score signifies a higher priority for enrollment. Veterans in priority group 5 are unique in that they're eligibility is based not on disability, but on income status (i.e. Medicaid eligibility).
Time Frame: 8 weeks
Population: VA Priority groups 4 & 5 only
Measure: Count of Participants; unit: Participants
Arm/Group | Screening | Awareness | Assistance
Number analyzed (Participants) | 43 | 48 | 52
Participants | 5 | 9 | 18
Statistical Analysis 1: Comparison: Screening; Test type: Superiority; p = 0.0094, Mixed Models Analysis; Odds Ratio (OR) = 5.006, 95% CI 2-sided [1.512 to 16.570], Standard Error of Mean 0.617 — This analysis is arm 1 compared to compared to arm 3. Arm 3 is the numerator and arm 1 is denominator
Statistical Analysis 2: Comparison: Screening; Test type: Superiority; p = 0.3377, Mixed Models Analysis; Odds Ratio (OR) = 1.875, 95% CI 2-sided [0.521 to 6.746], Standard Error of Mean 0.6532 — This is a comparison of arm 1 and arm 2. Arm 2 is the numerator and arm 1 is the denominator

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for 1 year for each participant from index screen to 12 months after.
Arm/Group | Screening | Awareness | Assistance
All-Cause Mortality (participants affected / at risk) | 5/161 | 3/160 | 2/158
Serious Adverse Events (participants affected / at risk) | 0/161 | 0/160 | 0/158
Other Adverse Events (participants affected / at risk) | 0/161 | 0/160 | 0/158

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/83/NCT04977583/Prot_SAP_001.pdf
  • Informed Consent Form (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT04977583/ICF_000.pdf